CLINICAL TRIAL: NCT07308821
Title: Effects of a Peer-mentoring Program on Undergraduate Students' Outcomes and Perspectives Related to a Career in Communication Sciences and Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY25-26-4917
Record Dates: First submitted 2025-12-09; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mentoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mentor group (Experimental)
  Interventions: Behavioral: mentor program
- comparison group (No Intervention)

INTERVENTIONS:
Behavioral: mentor program — mentor program participant
  Arms: mentor group

SUMMARY:
The purpose of the study is to investigate the effects of implementing a semester-long mentoring program in Communication Sciences & Disorders on its participants and how the experience differs from the students who did not participate.

DETAILED DESCRIPTION:
Speech-language pathology (SLP) and audiology (AUD) comprise the fields of communication sciences and disorders (CSD) and have consistently been considered professions both in-demand and facing job shortages. Speech-language pathology is facing a projected growth of 18 percent from 2023 to 2033 as a result of the increasing needs of the adult and pediatric populations with communication disorders that SLPs serve (American Speech- Language-Hearing Association [ASHA], n.d.). Similarly, the field of audiology is expected to continue expanding at an albeit smaller increase of 11 percent, but one that will be adding an average of 1,600 jobs a year to a market in need of qualified audiologists who often work alongside SLPs to provide services to those in need (ASHA, n.d.). This demonstrates positive growth and expansion of the field of SLP and AUD, but the job vacancies unfortunately outnumber the amount of job seekers available to assist these vulnerable populations and bolster the current SLP and AUD workforce (ASHA, 2024; ASHA, 2025). The discrepancy between the demand for SLPs/AUDs and the supply of qualified clinicians ready to enter the workforce has prompted a call to action (Castro, 2025). For this reason, research into how to best support undergraduate students who may one day be the future clinicians of tomorrow is an important focus area.

One such method of support is peer mentorship designed to assist students with becoming acclimated to their academic environment and creating robust social support networks that help them develop a sense of belonging and navigate the transition into higher education (Hall & Jaugietis, 2011; Rayle & Chung, 2007). Peer mentoring programs may also create supportive environments that help undergraduate students reduce the risk of school attrition, improve academic achievement, and foster social and professional skill development (Goff, 2011; Jacobi, 1991; Mahendra & Kashinath, 2022).

This study will be part of an ongoing process to understand how to increase interest in the SLP/AUD fields amongst undergraduate students and how to encourage the desire to pursue a graduate degree and eventually join the workforce that is in need of qualified CSD professionals.

ELIGIBILITY:
Inclusion Criteria: enrolled in CSND 100 -

Exclusion Criteria: not enrolled in CSND 100

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mentorship experiences survey developed by the research team | prestest at baseline (Feb 2026); immediately after completion of mentor program (May 2026)
  pre/post program survey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rayle, A. D., & Chung, K.-Y. (2007). Revisiting first-year college students' mattering: Social support, academic stress.Student Retention: Research, Theory & Practice, 9(1), 21-37. https://doi.org/10.2190/ x126-5606-4g36-8132
- [Background] Montclair State University. (2024, September 7). What It Means to Be a Hispanic-Serving University.https://www.montlcair.edu
- [Background] Mahendra N, Kashinath S. Mentoring Underrepresented Students in Speech-Language Pathology: Effects of Didactic Training, Leadership Development, and Research Engagement. Am J Speech Lang Pathol. 2022 Mar 10;31(2):527-538. doi: 10.1044/2021_AJSLP-21-00018. Epub 2021 Nov 3. PMID 34731580
- [Background] Jacobi, M. (1991). Mentoring and undergraduate academic success: A literature review. Review of Educational Research
- [Background] Hall, R., & Jaugietis, Z. (2011). Developing peer mentoring through evaluation. Innovative Higher Education, 36, 41-52. https://doi.org/10.1007/s10755-010-9156-6
- [Background] Goff, L. (2011). Evaluating the outcomes of a peer-mentoring program for students transitioning to postsecondary eTeaching and Learning, 2(2), Article 2. https://doi.org/10.5206/cjsotl-rcacea.2011.2.2
- [Background] Castro, N. (2025). Opening the pipeline to the field of communication sciences and disorders through career counseling 1-18. https://doi.org/10.1044/2025_PERSP-24-00291
- [Background] American Speech-Language-Hearing Association [ASHA]. (2025). Supply and demand resource list for audiologists audiologistshttps://www.asha.org/siteassets/surveys/supply-demand-audiology.pdf?srsltid=AfmBOooHaoNWkJCjuBfAtry3Yx9P
- [Background] American Speech-Language-Hearing Association [ASHA]. (2024). Schools survey report: SLP workforce and work for speech language pathologists chttps://www.asha.org/siteassets/surveys/schools-survey-report-slp-workforce-trends-2004-2024.pdf?srsltid=AfmBO
- [Background] American Speech-Language-Hearing Association [ASHA]. (n.d.). Market Trends in Audiology and Speech-Languaghttps://www.asha.org/careers/market-trends/#:~:text=audiologists%20and%20SLPs.-,Reasons%20for%20Growth,o